CLINICAL TRIAL: NCT06175806
Title: Oral Granisetron Versus Oral Ondansetron for Treatment of Gastroenteritis: A Randomized Controlled Clinical Trial
Brief Title: Granisetron Versus Ondansetron for Nausea and Vomiting in Pediatric Age Group
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ain Shams University (Other)
Responsible Party: Principal Investigator, Haya Essam Ibrahim, lecturer of pediatrics, Ain Shams University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: FMASU MS 519/2023
Record Dates: First submitted 2023-12-01; First posted 2023-12-19 (Actual); Last update posted 2023-12-19 (Actual); Status verified 2023-12

CONDITIONS: Nausea and Vomiting in Pediatric Age Group
MeSH Terms: conditions — Nausea

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- arm I (group A) who will receive dispersible film ondansetron (Experimental): arm I (group A) who will receive dispersible film ondansetron in a dose of 4 mg for those who will weigh more than 15 Kg up to 30 kg, and 8 mg for those who will weigh more than 30 Kg. The dose will be repeated if the patient had another vomiting episode within 15 minutes of taking the medicine.
  Interventions: Drug: Ondansetron Oral Film
- Arm II (group B) who will receive oral Granisetron (Experimental): Arm II (group B) who will receive oral Granisetron in a dose of 40 microgram/kg/dose; the dose could be repeated if needed after 12 hours.
  Interventions: Drug: Granisetron Oral Liquid Product

INTERVENTIONS:
Drug: Ondansetron Oral Film — 5-hydroxytryptamine (5-HT) receptor antagonist
  Arms: arm I (group A) who will receive dispersible film ondansetron
Drug: Granisetron Oral Liquid Product — 5-hydroxytryptamine (5-HT) receptor antagonist
  Arms: Arm II (group B) who will receive oral Granisetron

SUMMARY:
The current clinical trial will include 160 children who will be presented with vomiting to the Outpatient Department of the Children's Hospital, Faculty of Medicine, Ain Shams University. Participants will be assigned randomly to receive either a dispersible film Ondansetron or oral Granisetron. After initial assessment, both groups will be followed up after 6 and 48 hours to check the frequency of vomiting, diarrhea, fever, headache as well as the return of appetite and the need for further treatment. The impact of nausea and vomiting on patients' daily lives will be assessed using a modified version of the Functional Living Index-Emesis (FLIE).

ELIGIBILITY:
Inclusion Criteria:

• Patients presenting with vomiting within the past 24 hours, including patients without dehydration and those who have mild to moderate dehydration.

Exclusion Criteria:

* Patients who are severely dehydrated.
* Patients who have bloody vomiting.
* Children with chronic diseases like type 1 diabetes mellitus, end stage renal disease and who are receiving chemotherapy.
* Patients who have vomiting due to surgical causes like intestinal obstruction.

Ages: 4 Years to 14 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 160 (Actual)
Dates: Start 2023-09-10 (Actual); Primary Completion 2023-11-11 (Actual); Study Completion 2023-11-11 (Actual)

PRIMARY OUTCOMES:
To compare the effectiveness of Granisetron oral solution and Ondansetron oral dispersible film for treatment of vomiting in pediatric patients. | at 6 hours and at 48 hours of adminsteration
  The number of vomiting episodes.

CONTACTS AND LOCATIONS:
Overall Officials: Mohamed F Allam, MD, Principal Investigator — Professor of Family Medicine, Faculty of Medicine, Ain shams University; May F Nassar, MD, Study Director — Professor of pediatrics, Faculty of Medicine, Ain shams University; Ehab K Emam, MD, Study Chair — Professor of pediatrics, Faculty of Medicine, Ain shams University; Haya E Ibrahim, MD, Principal Investigator — lecturer of pediatrics,Faculty of Medicine, Ain shams University
Locations (1):
- Faculty of Medicine-Ain Shams University, Cairo, Abbasia, Egypt

IPD SHARING:
Plan to Share IPD: No